CLINICAL TRIAL: NCT00512460
Title: A Phase I Safety and Pharmacokinetic Study of Intravenous RTA 744 Injection in Patients With Recurrent, Progressive or Refractory Neoplastic Meningitis
Brief Title: RTA 744 Injection in Patients With Leptomeningeal Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was closed due to loss of industry sponsorship
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Reata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0506
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Neoplastic Meningitis; Solid Tumor; Lymphoma; Leukemia; Brain Tumor
Keywords: Neoplastic Meningitis; Leptomeningeal Disease; Solid Tumor; Lymphoma; Leukemia; Brain Tumor; RTA 744
MeSH Terms: conditions — Meningeal Carcinomatosis; Lymphoma; Leukemia; Brain Neoplasms; Meningeal Neoplasms | interventions — WP 744

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RTA 744 (Experimental)
  Interventions: Drug: RTA 744

INTERVENTIONS:
Drug: RTA 744 — 4.8 mg/m^2 by vein Over 2 Hours On Days 1-3.

SUMMARY:
1. The primary objectives of this study are:

   1. To determine the tolerability of RTA 744 Injection in patients with leptomeningeal disease (LMD) secondary to any type of primary tumor.
   2. In a selected group of 6-10 patients who will receive RTA 744 at or near the maximum tolerated dose (MTD), to characterize the multiple-dose pharmacokinetics of RTA 744 in plasma and CSF.
2. The secondary objectives of this study are:

   1. To document any potential antitumor activity of RTA 744 in this patient population.
   2. To correlate pharmacokinetic information with clinical (efficacy and safety) responses, as a possible help in selecting appropriate doses for later studies.

DETAILED DESCRIPTION:
RTA 744 is designed to enter the spinal fluid and kill cancer cells both in the spinal fluid and in the rest of body.

Before you can start receiving the study drug, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded. You will be asked about any drugs you have taken and are taking. You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). You will have a neurological exam. Blood (about 2 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative. Urine will be collected over a 24-hour period to test kidney function and for routine tests. You will have a magnetic resonance imaging (MRI) scan of the brain and spine.

You will have a chest x-ray. You will be asked questions about your ability to perform daily activities (performance status evaluation). You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will have either a multiple gated acquisition scan (MUGA) or an echocardiogram to check your heart's health. Samples (1 1/2 teaspoons) of cerebrospinal fluid from your spine and brain will be collected to look for the presence of cancer cells. The spinal sample will be collected through a lumbar puncture (spinal tap). The other sample will be taken from your brain through an Ommaya Reservoir tap. Radioactive dye will be injected into the CSF to make sure the CSF flows freely throughout the spinal canal. This is called an Indium-111 DPTA or Technetium 99m-DPTA Flow Study.

If you are found to be eligible to take part in this study, you should receive the same dose of RTA 744 throughout the study. The amount of study drug you receive will be determined by when you begin the study. Every 21 days on study is considered 1 study "cycle." If you have intolerable side effects, the drug dosing for the next cycle may be delayed for up to 21 days to allow any symptoms or side effects to resolve. You may be given a lower dose level.

The first participant on this study will receive the dose that has been found to be well-tolerated in an ongoing study involving participants with primary brain tumors. After this participant has completed 1 study cycle, the next participant will be given a higher dose of RTA 744. Each new participant will receive a higher dose level until a patient has an intolerable side effect. When this happens, at least 2 more participants will be given the dose level that causes the intolerable side effect. If there are no further intolerable side effects to RTA 744, the next group of 3 participants will be given the next higher dose of RTA 744. Each time, the dose of RTA 744 will not be increased until the effects of the previous dose level have been studied. Doses will increase with each group of patients until the highest tolerable dose is found.

On Day 1 Cycle 1, before you receive the first dose of RTA 744, you will have a physical exam, neurological exam, and a performance status evaluation. If the screening neurological exam was performed less than 1 week before Day 1, the neurological exam will not need to be repeated. You will also be asked about any drugs, treatments, or herbal medicines you are taking. You will be asked how you are feeling and if whether you are experiencing any symptoms or side effects. Blood (less than 2 tablespoons) and urine will be collected for routine tests, unless blood and urine were collected for screening within the past 72 hours.

After completion of these tests, you will receive RTA 744 through a needle in your vein over a 2-hour period on Days 1-3. You must remain in the clinic for 2 hours after the drug is given to make sure you are not having any side effects.

During Cycle 1, you will be asked to return to the clinic once a week for 3 weeks. At these visits, blood (less than 2 tablespoons) will be drawn for routine tests. You will be asked how you are feeling and whether you are having any side effects.

On Day 21, you will have a neurologic exam.

Before receiving the study drug on Day 1 of Cycles 2-18, you will have a physical exam, neurological exam, and a performance status evaluation. You will also be asked about any drugs, treatments, or herbal medicines you are taking. Blood (less than 2 tablespoons) and urine will be collected for routine tests. You will have an ECG. Before Cycles 4, 6, 8, 10, 12, 14,16, and 18, you will have a MUGA scan or an echocardiogram. Once you have completed the tests, you will receive the study drug in the same manner as Cycle 1.

During Days 1-3, you will be asked how you are feeling and to report any symptoms or side effects you may have noticed during or after receiving RTA 744.

On Day 15, blood (about 3 teaspoons) will be drawn for routine tests. This blood draw may be performed by an outside laboratory. If no clinic visit is scheduled on Day 15, you will be contacted by telephone to find out if you have experienced any side effects. This phone call should last less than 5 minutes.

On Day 21, blood (less than 2 tablespoons) will be drawn for routine tests.

One time (per cycle) between Day 15 and Day 21 of Cycles 2, 4, 6, 8, 10, 12, 14, 16, and 18, a sample (about 2 teaspoon each time) of CSF will be collected from your spine through a spinal tap, and from your brain through an Ommaya Reservoir tap. This will be done in order to look for cancer cells. You will also have an MRI of the brain and spine.

An ECG will be performed during the last week of all cycles. A MUGA scan or an echocardiogram will be performed during the last week of Cycles 4, 6, 8, 10, 12, 14, 16, and 18.

You will have an MRI within 1 week of the end of the last cycle.

You may remain on study for up to 18 cycles (13 months). You will be taken off study if the disease gets worse or intolerable side effects occur.

Once you are off study, you will have an end-of-study visit. At this visit, your complete medical history will be recorded. You will be asked about any drugs you have taken and are taking. You will have a physical exam, including measurement of vital signs. You will have a neurological exam. Blood (about 2 tablespoons) will be drawn for routine tests. Urine will be collected over a 24-hour period to test kidney function and for routine tests. You will have an MRI of the brain and spine.

You will have a chest x-ray. You will have a performance status evaluation. You will have ECG and MUGA scans or echocardiogram. Samples (1 1/2 teaspoons each) of cerebrospinal fluid from your spine and brain will be collected to look for the presence of cancer cells. The spinal sample will be collected through a spinal tap. The other sample will be taken from your brain through an Ommaya Reservoir tap. Radioactive dye will also be injected into the CSF to make sure the CSF flows freely throughout the spinal canal.

THIS IS AN INVESTIGATIONAL STUDY. RTA 744 is not FDA approved or commercially available. It has been authorized for use in research only.

Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18 years.
2. Histologic confirmation of primary malignancy at original diagnosis. All primary tumor types may be enrolled into the study (solid tumor, lymphoma, leukemia, or brain malignancy).
3. Neoplastic meningitis/leptomeningeal metastasis refractory to conventional intrathecal therapy and defined as presence of tumor cells on cytology after cytospin, OR neuroimaging evidence of leptomeningeal tumor by MRI accompanied by clinical evidence of leptomeningeal tumor.
4. Patient is not eligible for higher priority clinical trial.
5. If patient had surgical resection prior to enrollment, at least 2 weeks should have elapsed prior to enrollment into the study and patient must have completely recovered from the side effects of such therapy.
6. For those patients taking steroid medications, the dose of steroid should be stable for at least 7 days prior to obtaining the Gd-MRI of the brain and spine, if medically feasible.
7. Karnofsky Performance Status (KPS) of >/= 60.
8. Laboratory Parameters: 1) Absolute Neutrophil Count (ANC) >/=1.5 x 10^9/L; 2) Hemoglobin (Hgb) >/=9 g/dl; 3) Platelets >/= 100 x 10^9/L; 4) AST and ALT </= 3.0 x Upper Limit of Normal (ULN); 5) Serum bilirubin </= 1.5 x ULN; 6) Serum creatinine </= 1.5 x ULN and 24 hour creatinine clearance >/= 50 ml/min
9. Life expectancy of at least 8 weeks based on the judgment of the clinical investigator.
10. Written informed consent obtained.

Exclusion Criteria:

1. Concurrent intrathecal or intraventricular therapy for leptomeningeal disease or other malignancy.
2. Concurrent oral or intravenous cytotoxic therapy for leptomeningeal disease or other malignancy. Patients who are receiving non-cytotoxic concurrent drug for their malignancy may be allowed on the study, provided that the non-cytotoxic drug was started for at least 4 weeks prior to entry into the study and that no apparent toxicity from the non-cytotoxic drug is evident.
3. Clinical evidence of obstructive hydrocephalus or compartmentalization of CSF flow.
4. Patient has previously received anthracycline therapy up to the following cumulative doses: doxorubicin >/= 550 mg/m^2 (>/= 450 mg/m^2 if patient has had prior chest radiotherapy), epirubicin >/= 1000 mg/m^2 (>/= 800 mg/m^2 if prior chest radiation), idarubicin >/= 150 mg/m^2 (>/= 130 mg/m^2 if prior chest radiotherapy) and daunorubicin >/= 550 mg/m^2 (>/= 400 mg/m^2 if prior chest radiotherapy).
5. Patients on anticonvulsant medications or other types of medications which are known liver-enzyme inducers.
6. Patients who are pregnant or breast feeding, or adults (male or female) of reproductive potential not employing an effective method of birth control (such as oral, implantable, or injectable contraceptives ) (Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to administration of RTA 744 Injection)
7. Total urinary protein in 24 hours urine collection > 500 mg
8. Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study: 1) Uncontrolled diabetes (patients diagnosed with Type 1 or Type 2 diabetes who are currently under treatment by a physician for this condition and are not able to control blood sugars with management for glucose levels above 250 mg/dL). 2) Active or uncontrolled infection. 3) Acute or chronic liver disease (i.e., hepatitis, cirrhosis). 4) Confirmed diagnosis of HIV infection
9. Impaired cardiac function, other significant prior cardiac disease or arrhythmia of any type, including any of the following: 1) LVEF < 45% as determined by MUGA scan or echocardiogram. 2) Complete left bundle branch block. 3) Obligate use of a cardiac pacemaker. 4) ST depression of > 1mm in >/= 2 leads and/or T wave inversions in >/= 2 contiguous leads. 5) Congenital long QT syndrome.
10. 9. (continued) 6) History or presence of ventricular or atrial tachyarrhythmias. 7) Clinically significant resting bradycardia (< 50 beats per minute). 8) QTc > 480 msec on screening ECG. 9) Uncontrolled high blood pressure(>140/90), history of labile hypertension, or history of poor compliance with an antihypertensive regimen. 10) Unstable angina pectoris. 11) Symptomatic congestive heart failure.
11. Myocardial infarction </=6 months prior to starting study drug. Patients with a history of CHF or arrhythmias
12. Patients who are taking therapeutic doses of anticoagulant therapy (prophylactic dosing is allowed.)
13. Patients who have received the following types of prior or concurrent therapy, or who have not recovered from the toxic effects of such therapy: 1) investigational drugs less than 4 weeks prior to entry on this study. 2) intrathecal chemotherapy within 2 weeks prior to entry into this study. 3) systemic cytotoxic chemotherapy within 4 weeks prior (6 weeks for nitrosourea or mitomycin-C or 2 weeks for vincristine) to entry on this study. 4) radiation therapy within 2 weeks prior to entry on this study. 5) any medication known to cause QT interval prolongation.
14. Patients who have had any surgery, including resection of a brain tumor within 2 weeks prior to entry on this study
15. Patients unwilling to or unable to comply with the protocol
16. Patients who have a contraindication to MRI imaging (cardiac pacemaker, other ferromagnetic metal implants, claustrophobia not amenable to conscious sedation, and obesity greater than 300 lbs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To study the highest tolerable dose of RTA 744 that can be given to patients with cancer that has spread to the meninges of the brain or the spine. | 3 Years

SECONDARY OUTCOMES:
To study the level of effectiveness of RTA 744 on the disease. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Groves, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org